CLINICAL TRIAL: NCT01687140
Title: The Use of D-Cycloserine to Augment Intensive Cognitive Behavioral Therapy for Pediatric Obsessive Compulsive Disorder
Brief Title: The Use of D-Cycloserine to Augment CBT for Pediatric OCD
Acronym: DCS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, R. Lindsey Bergman, Principle Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NCT003135
Record Dates: First submitted 2012-09-13; First posted 2012-09-18 (Estimated); Last update posted 2012-09-18 (Estimated); Status verified 2012-09

CONDITIONS: Obsessive-Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Cycloserine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Participant takes one pill of placebo a day 4 times weekly immediately preceding the treatment session for two weeks of treatment (4 sessions weekly).
  Interventions: Drug: Placebo
- DCS (Active Comparator): Participant takes one pill of D-Cycloserine a day 4 times weekly immediately preceding the treatment session for two weeks of treatment (4 sessions weekly).
  Interventions: Drug: D-Cycloserine

INTERVENTIONS:
Drug: D-Cycloserine — Take one pill a day 4 times weekly immediately preceding the treatment session for two weeks of treatment (4 sessions weekly).
  Arms: DCS
Drug: Placebo — Take one pill a day 4 times weekly immediately preceding the treatment session for two weeks of treatment (4 sessions weekly).
  Arms: Placebo

SUMMARY:
Pediatric obsessive compulsive disorder (OCD) is a relatively common and often severe condition that can become chronic if untreated. One of the most effective treatments for OCD is a type of cognitive behavioral therapy called exposure and response prevention (ERP). ERP involves presenting a patient with feared objects or situations (the content of their obsessional fears) in a gradual manner while helping them use coping techniques to refrain from engaging in rituals (compulsions). Despite several studies suggesting that ERP is an effective treatment for pediatric OCD, many youngsters fail to respond to this treatment, or respond only partially.

An exciting recent finding from animal research is the ability of an established antibiotic (traditionally used to treat Tuberculosis), D-cycloserine (trade name: Seromycin) to enhance certain types of learning among rats. The type of learning that is enhanced is called extinction learning and many researchers believe that extinction learning is the equivalent process to what occurs during ERP; it is the process whereby repeated exposure to the object of fear without any bad outcome causes the object to cease being associated with danger. Several clinical trials using ERP and other forms of exposure treatment for adults with anxiety disorders reproduced this finding from the animal literature; pairing DCS with exposure treatment (comparable to extinction learning) resulted in greater fear reduction than when no DCS was administered. The effects of DCS on exposure treatment for anxiety disorders among children has been tested only preliminarily in one study of children with OCD and results were unclear with children who received DCS augmentation showing non-significant but increased levels of improvement as compared with children who did not receive DCS augmentation.

In this study, 26 youngsters ages 7-17 with a primary diagnosis of OCD will be recruited and assigned at random to one of the two treatment conditions. Youth in the DCS condition of the study will receive 50 mg DCS 1 hr prior to each treatment session, while youth in the placebo condition receive an identical placebo capsule 1 hr prior to each treatment augmentation session. All participants will receive 180 minutes of CBT for OCD 4 days per week for 2 weeks during their study participation (as included in IOP already). All families complete a thorough evaluation no more than 5 days prior to receiving DCS on their 9th treatment visit in IOP (third week), and at mid-treatment augmentation (after the 12th IOP treatment session), post-treatment augmentation (after the 16th IOP treatment session), and 3-month follow-up (12 weeks after the 16th IOP treatment session). The primary aim of this study is to obtain preliminary data comparing the effects of the acute administration of DCS versus placebo on symptom response to exposure treatment for pediatric OCD. Results from this study will help to inform and refine future studies, and eventually, impact treatments for pediatric OCD.

DETAILED DESCRIPTION:
Although research has demonstrated clear benefits of cognitive behavioral treatment for children with obsessive-compulsive disorder, typical rates of treatment response are far from absolute and even treatment responders tend to exhibit continuing symptoms. In one of the most cited and largest child OCD treatment study to date, only 39% of the participants showed a robust response to a 12-week course of CBT. In recent years, the basic research finding that D-Cyclocerine, a partial N-methyl-Daspartate (NMDA) receptor agonist, enhances extinction of learned fear among rats2 has generated significant interest among clinical researchers. This is not surprising given that the core component of CBT involves exposing the individual to the feared stimuli in the absence of the feared consequence (ie, extinction training). Indeed, data from several trials (for adults with social anxiety, specific phobia, and OCD) indicate that compared to placebo, when DCS is added to exposure, participants tend to respond faster and at higher rates to treatment. This significant development in clinical treatment for anxiety disorders has been examined in only one pilot study among children with OCD. In this study, the effects of DCS were modest but the methodology utilized (eg., no objective symptom measure, lack of information regarding aspects of treatment) make the results difficult to interpret. The present study will help clarify, albeit in only a preliminary way, whether DCS is a promising addition to the treatment options available to the OCD treatment provider. The greatest utility of the augmentation strategy may be the capability to hasten the rate of improvement, and thus, decrease the discomfort of treatment and decrease treatment drop-out.

*Research Design and Methods: Describe in detail the design and methodology of the study.

A) Overview We propose to examine the preliminary efficacy of D-cycloserine augmentation of eight sessions (two weeks) of intensive exposure and response prevention treatment administered to youngsters aged 7-17 with primary OCD. All subjects will be receiving clinical treatment through the UCLA Child OCD Intensive Outpatient Program and DCS will be introduced, and will be delivered during the third and fourth week (starting on the 9th IOP treatment visit) of the subject's participation in the IOP clinical treatment.

To best address these aims, a total twenty-six 7-17 year-old children and adolescents will be recruited from UCLA Child OCD Intensive Outpatient Program. After completing an eligibility screen, all qualified participants will undergo a baseline evaluation including diagnostic as well as symptom assessments before randomization or treatment. This baseline assessment will be completed no more than 5 days prior to their 9th treatment visit (i.e., their first day of DCS medication).

Following these assessments, subjects will be randomized to receive either DCS or placebo (PBO) 4 times weekly immediately preceding their treatment session for two weeks of treatment (4 sessions weekly). Study participants will receive the same cognitive-behavior treatment through IOP whether they are in the active (DCS) or placebo (PBO) condition. In addition, all subjects will continue clinical treatment in IOP for as long as clinically indicated. However, responders at study week 2 (CGI-I = 1 or 2) will be reassessed at three-month follow-up to establish durability of early response. Parents will participate in the child's clinical assessment, and fill out self-reports, to better help the research team understand the child's functioning. Please see attached table of procedures for overview.

B. Core Clinical Assessment (Visit 1):

Diagnostic assessment will be based on the Anxiety Disorder Interview Schedule for DSM-IV, Child Version and Parent Version (ADIS-C & ADIS-P; Silverman & Albano, 1996). The ADIS is a structured interview schedule designed to obtain information about symptomatology, course, etiology, and severity of anxiety disorders, mood disorders, and externalizing disorders in children and adolescents. The following sections will be administered at this visit: all anxiety disorders (except selective mutism), anxiety disorder NOS, MDD, dysthmia, bipolar, ADHD, CD, ODD, substance use disorders, and tic disorders. The ADIS currently provides the basis for psychiatric diagnosis in our ongoing CAMELS Study for which the Child OCD, Anxiety, & TS program is a collaborating center. All potential research subjects will undergo ADIS assessment by one of the trained study clinical interviewers. The ADIS interview will take approximately 90 minutes to complete and will be administered only at baseline.

All study subjects will complete a core battery of dimensional psychiatric rating scales to more fully characterize OCD along with other key variables, including demographic status, other comorbid symptomatology, functional status, and adverse events or side effects. Many of these measures are derived from recent or ongoing treatment protocols in our OCD, Anxiety and Tic Disorders Program. In addition to the ADIS, the core battery will include the following measures:

1. Demographics/History. Provides standardized information regarding demographic status, medical history, and past history of mental health treatment. (10 minutes, only at baseline)
2. Children's Yale-Brown Obsessive Compulsive Scale (CY-BOCS): is a semi-structured clinical rating scale assessing OCD severity. The CY-BOCS was developed at Yale University for the definition of OCD symptoms and severity in children. The CY-BOCS will only be administered to youngsters with either parent- or child-report of obsessions or compulsions during the ADIS interview. (30 minutes at baseline administration; 15 minutes at end of study week 1, week 2, week 4, week 6, week 10, and 3-month follow-up)
3. Child OCD Impact Scale Child OCD Impact Scale (COIS; Piacentini et al., 2003) is a reliable and valid self-report measure of OCD-related functional impairment. (5-10 minutes at baseline, end of study week 1, week 2, and 3-month follow-up).
4. Children's Depression Inventory - (Kovacs, 1992). The CDI is a psychometrically sound rating scale comprised of 27 items (rated 0-2) assessing depressive symptomatology over the preceding 2 weeks. Age and gender-based T-scores are generated for five factors of depression. (10 minutes at baseline, end of study week 2, and 3-month follow-up).
5. Clinical Global Impression of Severity (CGI-S): A clinician rated instrument designed to measure overall illness severity at that specific time point. This measure will be recorded at each time point but is clinician rated and will not affect subject burden.
6. Clinical Global Impression of Improvement (CGI-I): A clinician rated instrument designed to measure overall symptom improvement at that specific time point relative to baseline symptom severity. This measure will be recorded at each time point but is clinician rated and will not affect subject burden.
7. Side Effects and Adverse Events: Side effect and adverse events will be assessed at every visit using the using an amended Adverse Event Form from another study with which our group is involved. (5 minutes).
8. Behavioral Approach Test (BAT): We have adapted the BATs for this study from Ollendick et (2011) who developed BATs specifically for children. When possible, BATs will be realistic in that children will be asked to approach and/or touch actual feared object or situation. When that is not possible, children pictures or video will be used. BAT assessments will be designed idiographically for each participant based upon their responses to the clinician administered CYBOCS instrument. The task will be administered at baseline (study week 0), at end of study week 1, and end of treatment (end of study week 2). The BATs consisted of a series of gradually more difficult steps (ranging from 7 to 12 steps depending on the specific phobia). Due to the variability in number of steps on the BATs, percentage of steps completed will be used as the primary behavioral measure of BAT performance.

For the BAT, the child will be instructed to do their best, but also informed they can terminate the BAT at any time if they wish to do so. BATs are terminated at the child's request or when the terminal step is achieved. Children are asked to provide ratings of their anxiety utilizing SUDS ranging from 0 to 8 (0 = None, 2 = A Little, 4 = Some, 6 = A Lot, and 8 = Very Much). Ratings are obtained immediately following the last step of the BAT. (15-20 minutes at baseline, end of study week 1, end of study week 2, and 3-month follow-up).

Staff training and supervision on these and other project-specific clinical measures will be coordinated and supervised by senior research study personnel using standardized methods to maintain reliability over time. This portion of the assessment is estimated to take approximately 1.5 hours to 2 hours.

F. Procedure:

Following these assessments, a total of 26 eligible subjects from the UCLA IOP will be randomized by a computer-generated program in the UCLA research pharmacy in a double-blinded fashion to receive either eight-sessions of DCS augmented exposure plus response prevention (ERP +DCS) treatment (four times per week for 2 weeks) or eight sessions of placebo and ERP (ERP+PBO) for the same time period. All study staff and families have no knowledge of whether the individual youngsters are receiving placebo or DCS. All subjects will be clinically assessed after the first and second study weeks of treatment and again 12 weeks later. Additionally, there will be brief assessments (CY-BOCS and CGI measures) for the end of study weeks 4, 6, and 10. Parents will also participate in the child's clinical assessment, and fill out self-reports, to better help the research team understand the child's functioning. Please see attached table of procedures for overview.

ELIGIBILITY:
Inclusion Criteria:

* Ages 7 through 17 inclusive at the time of initial evaluation.
* Meets DSM-IV diagnostic criteria for OCD.
* Child is fluent English speaker.
* Parent Informed Consent and Child Informed Assent. Parents must agree to their child's participation in this protocol. Parents will be asked to fill out self-report questionnaires and participate in assessments that will provide us with more information about their child, however parents are not considered "participants" within this protocol, as all treatment is targeted toward their child.

Exclusion Criteria:

* IQ < 80 on the Wechsler Abbreviated Scale of Intelligence (WASI)
* Excessive or Problematic Substance Use or DSM-IV Conduct Disorder within the past 3 months.
* Lifetime DSM-IV diagnosis of PDD, Mania, or Psychotic Disorder.
* Any serious psychiatric, pscyhosocial, or neurological condition (i.e., ADHD, MDD, anxiety, severe aggression, family discord) requiring immediate treatment).
* Presence of primary hoarding symptoms or mental rituals.
* Having epilepsy, renal insufficiency, or generally poor physical health.
* Pregnancy or having unprotected sex (in females).

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Estimated)
Dates: Start 2012-07; Primary Completion 2014-07 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
OCD symptom severity on the Children's Yale Brown Obsessive Compulsive Scale (CYBOCS) | Post-treatment (Study day 9)
  Treatment outcome will be evaluated based on decreases in total OCD symptom severity as measured by the CYBOCS.

CONTACTS AND LOCATIONS:
Overall Officials: Lindsey Bergman, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States